CLINICAL TRIAL: NCT00004013
Title: Treatment of Refractory Stage IV Metastatic Breast Cancer With Weekly Paclitaxel or Weekly Paclitaxel and Herceptin Following Autologous/Syngeneic Stem Cell Transplant
Brief Title: Paclitaxel With or Without Trastuzumab Following Peripheral Stem Cell Transplantation in Treating Patients With Refractory Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1338.00; FHCRC-1338.00; GENENTECH-FHCRC-1338.00; NCI-G99-1557; CDR0000067230 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel

INTERVENTIONS:
Biological: trastuzumab
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Paclitaxel may stop the growth of breast cancer by stopping blood flow to the tumor.

PURPOSE: Phase II trial to compare the effectiveness of paclitaxel with or without trastuzumab following peripheral stem cell transplantation in treating patients who have refractory stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of paclitaxel with or without trastuzumab following high dose chemotherapy with autologous or syngeneic peripheral blood stem cell transplantation in patients with stage IV breast cancer. II. Assess the overall survival of these patients.

OUTLINE: Patients begin study treatment within 50-150 days after autologous or syngeneic peripheral blood stem cell transplantation. Patients are stratified according to overexpression of HER2-Neu (yes vs no), which determines the type of therapy. Arm I (overexpression of HER2-Neu): Patients receive paclitaxel IV over 60 minutes followed by the initial loading dose of trastuzumab IV over 90 minutes. If the loading dose is tolerated well, then patients receive maintenance trastuzumab IV over 30 minutes. Treatment with paclitaxel followed by maintenance trastuzumab repeats once every week for 12 weeks in the absence of disease progression or unacceptable toxicity. Arm II (no overexpression of Her2-Neu): Patients receive paclitaxel IV over 60 minutes once every week for 12 weeks. Patients with hormone receptor positive disease also receive antihormonal therapy (tamoxifen or anastrozole) as clinically indicated. Patients with isolated metastasis such as a single bone lesion may receive radiotherapy to that site after completion of study treatment. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients (30 per arm) will be accrued for this study over 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Refractory stage IV breast cancer Received high dose chemotherapy (HDC) with autologous or syngeneic peripheral blood stem cell transplantation (PBSCT) OR Stage IV breast cancer Failed to achieve complete response to HDC with autologous or syngeneic PBSCT at initial restaging following HDC No enrollment on protocol FHCRC-976, unless evidence of no response or progressive disease at initial restaging following transplantation Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Not specified Menopausal status: Not specified Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Platelet count at least 50,000/mm3 (untransfused) Absolute neutrophil count greater than 1,000/mm3 (without filgrastim (G-CSF) support) Hepatic: Bilirubin no greater than 2.5 times upper limit of normal (ULN) SGOT no greater than 2.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: LVEF greater than 40% No poorly controlled arrhythmias No prior coronary artery disease No congestive heart failure within last year No myocardial infarction within past 2 years Other: No active infection No grade 3 regimen related toxicity according to Bearman model No allergy to paclitaxel, trastuzumab, or benzyl alcohol No grade 3 peripheral neuropathy with last chemotherapy HIV negative Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics Endocrine therapy: Concurrent antihormonal therapy (tamoxifen or anastrozole) allowed as clinically indicated for hormone receptor positive disease Radiotherapy: Not specified Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1999-01; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona A. Holmberg, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States